CLINICAL TRIAL: NCT05801029
Title: A Phase II, Open-label, Single-arm, Multi-centre Study to Evaluate the Safety and Efficacy of Osimertinib With Amivantamab as First-line Treatment in Participants With Epidermal Growth Factor Receptor Mutation-Positive, Locally Advanced or Metastatic Non-small Cell Lung Cancer (OSTARA)
Brief Title: A Study to Investigate Safety and Efficacy of Osimertinib and Amivantamab in Participants With Non-small Cell Lung Cancer With Common Epidermal Growth Factor Receptor Mutations
Acronym: OSTARA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5162C00052
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; Non squamous; Epidermal Growth Factor Receptor (EGFR); Epidermal Growth Factor Receptor mutation (EGFRm)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib+Amivantamab (Experimental): Participants will receive osimertinib and amivantamab.
  Interventions: Drug: Osimertinib; Drug: Amivantamab

INTERVENTIONS:
Drug: Osimertinib — Osimertinib will be administered as 80 mg oral tablet once daily (from Day 2) until progression of disease or until a study intervention discontinuation criterion is met.
Drug: Amivantamab — Amivantamab will be administered as an IV infusion at 1050 mg (< 80 kg body weight) or 1400mg (≥ 80 kg body weight) (in 28-day cycles: once weekly in Cycle 1 (with a split dose on Days 1 to 2) and then every 2 weeks in subsequent cycles) until progression of disease or until a study intervention discontinuation criterion is met. The first cycle dose is spilt over 2 days- 350 mg on day 1 and 700 mg [body weight < 80 kg] or 1050 mg [body weight ≥ 80 kg] on day 2.

SUMMARY:
This study will assess the safety and efficacy of Osimertinib with Amivantamab as First-line Treatment in Participants with Epidermal Growth Factor Receptor Mutation-Positive, Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase II, open-label, single-arm, multi-centre study to assess the safety and efficacy of osimertinib with amivantamab as first-line treatment in adult participants with a local preexisting positive approved tissue test result for EGFRm (Ex19del or L858R), locally advanced (clinical stage IIIB, IIIC), metastatic (clinical stage IVA or IVB), or recurrent non-squamous NSCLC.

This study consists of screening period of 28 days, followed by the study intervention period wherein the participant receives treatment from Day 1 until disease progression or study intervention discontinuation. Participants will be followed up at week 6 (± 1 week), week 12 (± 1 week), then every 12 weeks (± 1 week) until radiological disease progression. Survival follow up will be performed every 12 weeks. Upon study intervention discontinuation a 28 day follow up visit will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented non-squamous NSCLC. NSCLC of mixed histology is allowed.
* Newly diagnosed locally advanced or metastatic NSCLC or recurrent non-squamous NSCLC, not amenable to curative surgery or radiotherapy.
* WHO PS of 0 to 1 with no deterioration over the 2 weeks prior to enrolment.
* Minimum life expectancy > 12 weeks at Day 1.
* Confirmation by the local laboratory that the tumour harbours one of the 2 common EGFRm known to be associated with (Epidermal Growth Factor Receptor- Tyrosine Kinase Inhibitor) EGFR-TKI sensitivity.
* At least 1 lesion that can be accurately measured at baseline as ≥10 mm in the longest diameter with computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurements.
* Contraceptive use by males or females should be consistent with local regulations

Exclusion Criteria:

* Any evidence of diseases, history of allogenic organ transplant, which in the investigator's opinion makes it undesirable for the participant to participate in the study or would jeopardise compliance with protocol.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the osimertinib, or previous significant bowel resection that would preclude adequate absorption distribution, metabolism, or excretion of osimertinib.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥2 years.
* Any unresolved toxicities from prior therapy with Common Terminology Criteria for Adverse Events CTCAE) Grade ≥1, at the time of first dose of study intervention, with the exception of alopecia and Grade 2 prior platinum therapy related neuropathy.
* Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring corticosteroids for at least 2 weeks prior to start of study intervention.
* Active infection, including tuberculosis and infections with HBV (verified by known positive HBsAg result) or HCV.
* Should participants with HIV infection be included, patients are only eligible if they meet the criteria per protocol.
* Patient with protocol defined cardiac issue.
* History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD.
* Any concomitant medications known to be associated with Torsade de Pointes.
* Prior exposure to any systemic anti-cancer therapy for advanced NSCLC not amenable to curative surgery or radiation including chemotherapy, biologic therapy, immunotherapy, or any investigational drug.
* Any concurrent anti-cancer treatment without an adequate washout period prior to the first dose of study intervention.
* Palliative radiotherapy with a limited field of radiation within 2 weeks, or with wide field of radiation or to more than 30% of the bone marrow within 4 weeks, prior to the first dose of study intervention.
* Major surgical procedure or significant traumatic injury.
* Current use of medications or herbal supplements known to be strong inducers of CYP 3A4.
* Prior treatment with an EGFR-TKI.
* Participants with a history of hypersensitivity, or intolerance to the active or inactive excipients of osimertinib, amivantamab, or recommended pre-treatments of amivantamab or drugs with a similar chemical structure or class to these drugs.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From screening (Day-28) to survival follow up (Approximately 52 months after the first participant is dosed)
  To assess the safety and tolerability of osimertinib plus amivantamab in participants with EGFR mutation-positive, locally advanced, or metastatic NSCLC.
Progression Free Survival (PFS) | From date of first dose of study intervention until radiological disease progression or death due to any cause (Approximately 52 months after the first participant is dosed)
  The time from date of first dose of study intervention until progression per RECIST 1.1 as assessed by the investigator at the local site, or death due to any cause. The analysis will include all dosed participants. All events will be included, regardless of whether the participant withdraws from therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of first dose of study intervention until death due to any cause. Landmarks at 18 and 24 months. (Approximately 52 months after the first participant is dosed)
  Time from date of first dose of study intervention until the date of death due to any cause. The analysis will include all dosed participants. All deaths will be included, regardless of whether the participant withdraws from therapy or receives another anti-cancer therapy.
Objective Response Rate (ORR) | From screening (Day -28) to radiological disease progression (Approximately 52 months after the first participant is dosed)
  The proportion of participants who have a confirmed complete response (CR) or confirmed partial response (PR), as determined by the investigator at local site per RECIST 1.1. The analysis will include all dosed participants with measurable disease at baseline.
Duration of Response (DoR) | From screening (Day -28) to radiological disease progression (Approximately 52 months after the first participant is dosed)
  The time from the date of first documented response until date of documented progression per RECIST 1.1 as assessed by the investigator at local site or death due to any cause. The analysis will include all dosed participants with measurable disease at baseline who have a confirmed response.

CONTACTS AND LOCATIONS:
Locations (20):
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Malaysia (5):
  - Research Site, George Town
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Kuching
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Yunlin
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home